CLINICAL TRIAL: NCT06627504
Title: Mechanisms Underlying the Relationship Between Sleep and Circadian Health and Cardiometabolic Risk in Adolescents With Type 1 Diabetes
Brief Title: Type 1 Diabetes REst for Metabolic Health
Acronym: T1DREaM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-1490; R01HL174735 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes (T1D); Sleep Health
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Health and Circadian Timing Intervention (Experimental): Participants will be prescribed a sleep schedule that allows them to obtain at least 1h more time in bed compared to their typical school week schedule. In addition, participants will be provided with pharmaceutical-grade exogenous melatonin and instructed to take 500mcg 2 hours before their scheduled bedtime. They will also be asked reduce evening light exposure starting 2 hours before bedtime by limiting household lights and dimming electronics. In the mornings, participants will be exposed to bright light for 30 minutes after waking by wearing provided ReTimer light therapy glasses.
  Interventions: Behavioral: Sleep Health and Circadian Timing Intervention
- Typical Sleep (No Intervention): Participants will be asked to sleep on their usual schedule.

INTERVENTIONS:
Behavioral: Sleep Health and Circadian Timing Intervention — Participants will be prescribed a sleep schedule that allows them to obtain at least 1h more time in bed compared to their typical school week schedule. In addition, participants will be provided with pharmaceutical-grade exogenous melatonin and instructed to take 500mcg 2 hours before their scheduled bedtime. They will also be asked reduce evening light exposure starting 2 hours before bedtime by limiting household lights and dimming electronics. In the mornings, participants will be exposed to bright light for 30 minutes after waking by wearing provided ReTimer light therapy glasses.
  Arms: Sleep Health and Circadian Timing Intervention

SUMMARY:
Research has shown a link between poor sleep health and late circadian timing with cardiometabolic health in adolescents with type 1 diabetes (T1D). Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in T1D, which begins as early as adolescence, and current therapies are limited. Therefore, this study plans to investigate whether cardiometabolic health can be improved with increased sleep duration and advanced circadian timing in adolescents with T1D with habitually insufficient sleep. To answer this question, investigators will study adolescents with T1D who get <7h sleep on school nights and measure changes in insulin sensitivity, glycemic control, and vascular function after one month of a sleep and circadian intervention (1+ hour longer time in bed each night plus evening melatonin and morning light therapy) compared to one month of typical sleep (usual school schedule).

ELIGIBILITY:
Inclusion Criteria:

* High school students between the ages of 14-19 years;
* Diagnosed with T1D for ≥1 year;
* Using an insulin pump or other automated insulin delivery system;
* Have typically insufficient sleep, defined by ≤ 7 h per night on school days (assessed by actigraphy);
* With or at risk for obesity based on either above-average weight (BMI ≥50th percentile) or parental history of obesity (BMI ≥ 30 kg/m2);
* Tanner stage 4 or 5, based on breast development for girls and testicular size for boys.

Exclusion Criteria:

* Prior diagnosis of a sleep disorder (e.g., insomnia, obstructive sleep apnea) or an elevated screening score on the OSA subscale of the Sleep Disorders Inventory for Students-Adolescents measure
* Regular use of medications affecting sleep (e.g., stimulants, atypical antipsychotics, melatonin or other sleep aids);
* Regular use of medications affecting IR (systemic steroids, adjunctive diabetes medications);
* HbA1c ≥12%;
* Severe illness or DKA within 60 days;
* IQ<70 or severe mental illness impacting sleep or ability to participate in the study;
* Night-shift employment or other obligations that would preclude adherence to the intervention.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | Baseline (following 1 month typical sleep) and following 1 month intervention
  Steady-state glucose infusion rate (M) normalized to free fat mass (FFM) and to steady-state insulin (M/I, [mg/kg FFM/min]/insulin) measured with hyperinsulinemic euglycemic clamp
Cardiovascular Function | Baseline (following 1 month typical sleep) and following 1 month intervention
  Value of central aortic stiffness from cardiovascular MRI
Glycemic Control | Baseline (following 1 month typical sleep) and following 1 month intervention
  Value of mean sensor glucose assessed with continuous glucose monitor

SECONDARY OUTCOMES:
Inflammation | Baseline (following 1 month typical sleep) and following 1 month intervention
  Laboratory values of hs-CRP, IL-6, and TNF-alpha
Adipokines | Baseline (following 1 month typical sleep) and following 1 month intervention
  Laboratory values of leptin and adiponectin
Cortisol | Baseline (following 1 month typical sleep) and following 1 month intervention
  Laboratory values of cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Simon, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All fully deidentified raw and processed/scored data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access to the data will be made at the end of the grant award or when a publication has been submitted. Once the data are submitted, the archive will control the long-term persistence of the data set.